CLINICAL TRIAL: NCT02105272
Title: Efficacy and Safety Study of OPC-1085EL Ophthalmic Solution in Subjects With Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1085EL-13-002
Record Dates: First submitted 2014-03-27; First posted 2014-04-07 (Estimated); Results first posted 2015-11-17 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-11

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- OPC-1085EL ophthalmic solution (Experimental): Once daily
  Interventions: Drug: OPC-1085EL ophthalmic solution
- Latanoprost ophthalmic solution (Active Comparator): Once daily
  Interventions: Drug: Latanoprost ophthalmic solution

INTERVENTIONS:
Drug: OPC-1085EL ophthalmic solution
  Arms: OPC-1085EL ophthalmic solution
Drug: Latanoprost ophthalmic solution
  Arms: Latanoprost ophthalmic solution

SUMMARY:
The purpose of this study is to determine the efficacy and safety of OPC-1085EL ophthalmic solution in comparison with latanoprost ophthalmic solution in subjects who are insufficiently responsive to latanoprost ophthalmic solution.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with diagnosis of bilateral primary open-angle glaucoma or ocular hypertension

Exclusion Criteria:

* Subjects with ocular conditions as defined by the protocol

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2014-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Kansai Region, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- OPC-1085EL Ophthalmic Solution: Once daily
  OPC-1085EL ophthalmic solution
- Latanoprost Ophthalmic Solution: Once daily
  Latanoprost ophthalmic solution
Period: Overall Study
Arm/Group | OPC-1085EL Ophthalmic Solution | Latanoprost Ophthalmic Solution
Started | 118 | 119
Completed | 113 | 116
Not Completed | 5 | 3
Not completed — Adverse Event | 1 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OPC-1085EL Ophthalmic Solution | Latanoprost Ophthalmic Solution | Total
Number analyzed (Participants) | 118 | 119 | 237
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 71 | 69 | 140
  >=65 years | 47 | 50 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (11.4) | 60.8 (11.5) | 60.4 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 76 | 137
  Male | 57 | 43 | 100
Region of Enrollment [Number; unit: participants]
  Japan | 118 | 119 | 237

OUTCOME MEASURES:

1. Primary Outcome: Decrease From Baseline in Intraocular Pressure
Time Frame: Baseline, week 8 predose
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | OPC-1085EL Ophthalmic Solution | Latanoprost Ophthalmic Solution
Number analyzed (Participants) | 117 | 118
mmHg | 2.9 [2.5 to 3.3] | 1.6 [1.2 to 2.0]

2. Secondary Outcome: Intraocular Pressure at Week 8 Predose
Description: Comparison of each group in intraocular pressure at Week 8 Predose. The number of subjects showed in the Participant Flow comes from all the subjects administered IMP. For efficacy analysis, on the other hand, several subjects were excluded from the analysis according to the statistical analysis plan. For example, subjects without IOP after administration were excluded. In addition, IOP measurement at 8 hours was not mandatory. That is why there are differences between the number in the Participant Flow and Outcome.
Time Frame: Week 8 Predose
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | OPC-1085EL Ophthalmic Solution | Latanoprost Ophthalmic Solution
Number analyzed (Participants) | 117 | 118
mmHg | 17.1 (0.2) | 18.4 (0.2)

3. Secondary Outcome: Intraocular Pressure at Week 8 at 2 Hours After IMP Administration
Description: Comparison of each group in intraocular pressure at Week 8 at 2 hours after IMP administration.
  The number of subjects showed in the Participant Flow comes from all the subjects administered IMP. For efficacy analysis, on the other hand, several subjects were excluded from the analysis according to the statistical analysis plan. For example, subjects without IOP after administration were excluded. In addition, IOP measurement at 8 hours was not mandatory. That is why there are differences between the number in the Participant Flow and Outcome.
Time Frame: Week 8 at 2 hours after IMP administration
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | OPC-1085EL Ophthalmic Solution | Latanoprost Ophthalmic Solution
Number analyzed (Participants) | 114 | 118
mmHg | 17.2 (0.2) | 18.2 (0.2)

4. Secondary Outcome: Intraocular Pressure at Week 8 at 8 Hours After IMP Administration
Description: Comparison of each group in intraocular pressure at Week 8 at 8hours after IMP administration.
  The number of subjects showed in the Participant Flow comes from all the subjects administered IMP. For efficacy analysis, on the other hand, several subjects were excluded from the analysis according to the statistical analysis plan. For example, subjects without IOP after administration were excluded. In addition, IOP measurement at 8 hours was not mandatory. That is why there are differences between the number in the Participant Flow and Outcome.
Time Frame: Week 8 at 8 hours after IMP administration
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | OPC-1085EL Ophthalmic Solution | Latanoprost Ophthalmic Solution
Number analyzed (Participants) | 88 | 92
mmHg | 16.7 (0.2) | 17.4 (0.2)

5. Secondary Outcome: Decrease From Baseline in Intraocular Pressure at Week 8 at 2 Hours After IMP Administration
Description: Comparison of each group in change from baseline in intraocular pressure at Week 8 at 2 hours after IMP administration.
  The number of subjects showed in the Participant Flow comes from all the subjects administered IMP. For efficacy analysis, on the other hand, several subjects were excluded from the analysis according to the statistical analysis plan. For example, subjects without IOP after administration were excluded. In addition, IOP measurement at 8 hours was not mandatory. That is why there are differences between the number in the Participant Flow and Outcome.
Time Frame: Baseline, Week 8 at 2 hours after IMP administration
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | OPC-1085EL Ophthalmic Solution | Latanoprost Ophthalmic Solution
Number analyzed (Participants) | 114 | 118
mmHg | 2.1 [1.7 to 2.4] | 1.0 [0.6 to 1.4]

6. Secondary Outcome: Decrease From Baseline in Intraocular Pressure at Week 8 at 8 Hours After IMP Administration
Description: Comparison of each group in change from baseline in intraocular pressure at 8 at 8 hours after IMP administration.
  The number of subjects showed in the Participant Flow comes from all the subjects administered IMP. For efficacy analysis, on the other hand, several subjects were excluded from the analysis according to the statistical analysis plan. For example, subjects without IOP after administration were excluded. In addition, IOP measurement at 8 hours was not mandatory. That is why there are differences between the number in the Participant Flow and Outcome.
Time Frame: Baseline, Week 8 at 8 hours after IMP administration
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | OPC-1085EL Ophthalmic Solution | Latanoprost Ophthalmic Solution
Number analyzed (Participants) | 88 | 92
mmHg | 1.7 [1.3 to 2.1] | 1.0 [0.6 to 1.3]

ADVERSE EVENTS:
Time Frame: From the start date of IMP administration to date of the final examination (up to Week 8 at e hours after IMP administration)
Arm/Group | OPC-1085EL Ophthalmic Solution | Latanoprost Ophthalmic Solution
Serious Adverse Events (participants affected / at risk) | 0/118 | 0/119
Other Adverse Events (participants affected / at risk) | 7/118 | 7/119
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OPC-1085EL Ophthalmic Solution (N=118) | Latanoprost Ophthalmic Solution (N=119)
Nasopharyngitis (Infections and infestations) | 4 (4) | 7 (8)
Glucose urine present (Investigations) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No